CLINICAL TRIAL: NCT02777710
Title: A Dose Escalation Phase I Study With an Extension Part Evaluating the Safety and Activity of an Anti-PDL1 Antibody (DURVALUMAB) Combined With a Small Molecule CSF-1R Tyrosine Kinase Inhibitor (PEXIDARTINIB) in Patients With Metastatic/Advanced Pancreatic or Colorectal Cancers
Brief Title: Evaluation of Safety and Activity of an Anti-PDL1 Antibody (DURVALUMAB) Combined With CSF-1R TKI (PEXIDARTINIB) in Patients With Metastatic/Advanced Pancreatic or Colorectal Cancers
Acronym: MEDIPLEX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: AstraZeneca (Industry); Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET15-037 (MEDIPLEX); 2015-002438-31 (EudraCT Number)
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — pexidartinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Pexidartinib-Durvalumab (Experimental): * DURVALUMAB (MEDI4736): therapeutic Class anti-PD-L1 mAb, given IV every 4 weeks at a fixed dose of 1500mg, AstraZeneca
  * PEXIDARTINIB (PLX3397): therapeutic Class Kinase inhibitor targeting CSF1-R, Flt3 and Kit. Administered daily as split dose regimen, orally. Five dose-levels possible in dose escalation part: 400mg 5 days on 2 days off (intermittent schedule), 400 mg, 600 mg, 800 mg or 1000 mg.
  In this combination trial, Pexidartinib should be taken first and the Durvalumab IV infusion should be scheduled 1 hour after the Pexidartinib morning dose.
  Interventions: Drug: Pexidartinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Pexidartinib — Treatment will be administered as long as patient experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent. If a DLT or a toxicity meeting the DLT definition but occurring outside of the DLT period, resolves to Grade ≤2 or the patient's baseline level within 14 days after toxicity onset, dosing may be resumed if agreed by the Sponsor at the same DL.
  Other Names: PLX3397
Drug: Durvalumab — Treatment will be administered as long as patient experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent. If a DLT or a toxicity meeting the DLT definition but occurring outside of the DLT period, resolves to Grade ≤2 or the patient's baseline level within 14 days after toxicity onset, dosing may be resumed if agreed by the Sponsor at the same DL.
  Other Names: MEDI4736

SUMMARY:
Colorectal cancer (CRC) and pancreatic ductal adenocarcinoma (PDAC) are the most common gastrointestinal cancers in Western countries and are both associated with significant morbidity and mortality. An intriguing similarity between CRC and PDAC is the fact that the newly developed immune checkpoint inhibitors, especially PD1/PDL1 inhibitors, seem to have limited efficacy as single agents in both of these tumor types. Recent preclinical studies point towards alternatively activated (M2-type) macrophages as possible culprits in inducing local immune protection from cytotoxic T cells and resistance to PD1/PD-L1 targeted agents. We hypothesize that CSF1R blockade will deplete the tumor microenvironment of M2 macrophages, thus favoring the induction of a cytotoxic anti-tumor T-cell response following PD-L1 blockade with an anti-PD-L1 monoclonal antibody. So we propose to conduct a Phase I dose escalation study in order to evaluate the safety and clinical activity of a combined treatment associating an anti-CSF1R (PEXIDARTINIB) with an anti-PD-L1 (DURVALUMAB) in patients with advanced/metastatic colorectal or pancreatic cancers. Dose escalation part will determine the Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of Pexidartinib given in combination with Durvalumab. Extension part will evaluate the clinical activity of the combination at the RP2D.

DETAILED DESCRIPTION:
This study will be a 2-part Phase I study comprising a dose-finding escalation part (to determine MTD/RP2D, safety and PK) followed by an extension part at RP2D. In the dose-escalation part, successive cohorts of 3 patients will receive Pexidartinib (given orally every day at escalating doses, five dose levels possible, Plexxikon), in combination with Durvalumab (given IV every 4 weeks at a fixed dose of 1500mg, AstraZeneca). The dose escalation scheme will be done using a Likelihood Continual Reassessment Method (CRML). After each new cohort of 3 patients is evaluated, model will be fitted and results will be discussed in a teleconference between the investigators, the sponsor, representatives of AstraZeneca and Plexxikon, and the statistician who will decide of the next dose to be assigned to the next cohort (Dose Escalation Meetings). In both parts, patients will continue to receive study drugs as long as they experience clinical benefit in the opinion of the investigator or until unacceptable toxicity including DLTs or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent. If a DLT or a toxicity meeting the DLT definition but occurring outside of the DLT period, resolves to Grade ≤2 or the patient's baseline level within 14 days after toxicity onset, dosing may be resumed if agreed by the Sponsor at the same DL. The extension part will comprise two independent cohorts of patients with pancreatic adenocarcinoma (PDAC cohort) or colorectal adenocarcinoma (CRC cohort) and biopsiable disease, and will allow the assessment of anti-tumor activity based on a Gehan design allowing to quickly identify treatments with low efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years at time of inform consent signature
* Histologically proven adenocarcinoma of the pancreas or colorectal, at the advanced or metastatic stage
* Prior therapy for the metastatic/advanced disease. For PDAC, treatment with at least one previous line of chemotherapy. For CRC, treatment with at least one previous line of therapy.
* Availability of a representative tumor specimen in paraffin blocks (preferred) or at least 20 unstained slides or a fresh tumor biopsy* before C1D1 with an associated pathology report. *: If there is no available archival material, a tumor biopsy has to be performed after patient' consent.
* Extension part: patients to be enrolled in this part of the study should have biopsiable disease (i.e. at least one lesion with a diameter of at least 10 mm, visible by medical imaging and accessible to percutaneous or endoscopic sampling)
* At least one measurable lesion according to RECIST 1.1
* ECOG PS 0-1
* Royal Marsden score of 0 or 1
* Adequate organ and marrow function as defined below based on medical records and according to lab tests performed within 72 hours before C1D1 (Hemoglobin ≥ 10.0 g/dL, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L; Lymphocyte count ≥ 0.5 x 109/L, Serum creatinine ≤ 1.5 × ULN and CL>60 mL/min using Cockcroft-Gault formula, or MDRD for patients over 65 years (Appendix 7- Creatinin clearance calculation), AST and ALT ≤ ULN, Serum bilirubin ≤ ULN (in the absence of Gilbert's syndrome), INR or PT ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy as long as INR/PT or PTT is within therapeutic range of intended use of anticoagulants, aPTT ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants, Serum potassium, magnesium, and calcium levels (high or low) ≤ Grade 1
* Minimal wash-out period for prior treatment (minimal time required from prior treatment and C1D1 of this study):Chemotherapy, immunotherapy, or radiation therapy > 14 days; Immunosuppressive medication > 28 days, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid; Live attenuated vaccination > 30 days; Strong CYP3A4 inducers or inhibitors > 14 days; Major surgical procedure, open biopsy (excluding skin cancer resection and screening tumor biopsy), or significant traumatic injury > 14 days (the wound must have healed).
* Women of child-bearing potential must have a negative serum pregnancy test within 72 hours before C1D1 and must agree to use 2 effective forms of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men must agree to use effective methods of birth control during the study and for up to 6 months after the last dose of study drug.
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Cancer disease considered curable with surgery or radiotherapy.
* Previous therapy with specific CTLA-4, CSF1, CSF1-R, PD-1 and/or PD-L1 inhibitors
* Persisting significant toxicities related to prior treatments i.e. ≥ Grade 2 AE according to CTCAE V4 except alopecia and biological values defined in inclusion criteria
* History of any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent,
* Inability to take oral medication (i.e. to swallow capsules of Pexidartinib) or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication.
* Hypersensitivity to the active substance or excipient or other humanized monoclonal antibody (a history of hypersensitivity reaction to cetuximab is allowed, but patient should be closely monitored for infusion-related reaction)
* Symptomatic or active leptomeningeal or parenchymal brain metastases. Patients with previously treated brain metastases (either by surgery, radiotherapy or radiosurgery) may be enrolled if stable, off steroids, on imaging and clinically, for at least 4 weeks.
* Active or prior/history of disease/medical condition listed below: Documented autoimmune disease within the past 2 years except for autoimmune hypothyroidism on a stable dose of thyroid supplementation and patients with type 1 diabetes mellitus on a stable dose of insulin. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded; Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction; Clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Patients must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months; Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis); Primary immunodeficiency; Allogeneic organ transplant; Known clinical diagnosis of tuberculosis; Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV); Any psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent; Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the sponsor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Patients with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible; hepatobiliary diseases including biliary tract diseases, autoimmune hepatitis, inflammation, fibrosis, cirrhosis of liver caused by viral, alcohol, or genetic reasons. Gilbert's disease is allowed if Total Bilirubine is ≤ 1.5 × ULN.
* Need for the following concomitant medications/interventions not permitted during the study treatment period: Any investigational anticancer therapy other than the protocol-specified therapies; Any concurrent chemotherapy, radiotherapy (except palliative radiotherapy on a non-target lesion after discussion with the sponsor), immunotherapy, biologic or hormonal therapy for cancer treatment, other than any stated in the protocol; Immunosuppressive medications including, but not limited to systemic corticosteroids at doses exceeding 10 mg/d of prednisone or equivalent, methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of investigational product-related AEs or in subjects with contrast allergies is acceptable; Live attenuated vaccines; Strong inhibitors and inducers of CYP3A4; Major surgery
* Pregnant or breast-feeding female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
part 1 (dose escalation part) : Dose-Limiting Toxicities (DLT) | during the DLT assessment window (i.e. 1 cycle = 28 days)
  A DLT is defined as one of the following toxicities occurring during the DLT assessment window (i.e. 1 cycle = 28 days) related to Durvalumab, Pexidartinib or both: any Grade ≥4 irAE, any Grade ≥3 irAE, that does not downgrade to Grade 2 within 3 days after onset of the event despite optimal medical management or does not downgrade to ≤ Grade 1 or baseline within 14 days, any Grade 2 pneumonitis that does not resolve to ≤ Grade 1 within 3 days of the initiation of maximal supportive care, Grade ≥ 4 neutropenia (ANC < 500/μL) lasting ≥ 7 days, Grade ≥ 3 febrile neutropenia, Grade ≥ 4 thrombocytopenia associated with clinically significant bleeding and lasting > 72 hours, AST/ALT > 10 x ULN, AST/ALT > 3x ULN with bilirubin >2x ULN, any other study drug related toxicity considered significant in the opinion of the investigators, any other Grade ≥ 3 major organ adverse event with some exceptions.
part 2 (extension part) : objective response rate (ORR) | 16 weeks of treatment
  The objective response rate (ORR) will be defined as the proportion of patients (described on the efficacy-evaluable population) who achieve complete response (CR) or partial response (PR) as best overall response at 16 weeks of treatment. ORR is based on tumor assessments (measurements according to RECIST 1.1 criteria).

SECONDARY OUTCOMES:
The duration of response (DoR) | from the time of first documented response (CR or PR as per RECIST 1.1 criteria) until the first documented progression or date of death due to underlying cancer, or censored at the date of the last available tumor assessment, assessed up to 52 weeks.
  in parts 1 and 2
Progression-Free Survival (PFS) | from the date of inclusion until the date of the first progression or date of death from any cause, up to 52 weeks.
  in parts 1 and 2, PFS will be estimated using the Kaplan-Meier method.
Adverse events reporting | from the signature of the ICF and the first intake of study drug until 90 days after the last study drugs intake or until initiation of a new anti-cancer treatment
  based mainly on the frequency of adverse events based on the common toxicity criteria (CTCAE-V4.03) grade.
Area under the Pexidartinib plasma concentration (AUC) versus time curve | Cycle 1 Day 1, C1D15, C2D1 and C3D1
  analyzed by measurement of area under the plasma concentration-time curve (AUC 0-4h, AUC 0-6h. For each time frame: at pre-dose of both study drugs and at 1, 2, 4 and 6 hours post- Pexidartinib dosing.
Peak Pexidartinib plasma concentration (Cmax) | Cycle 1 Day 1, C1D15, C2D1 and C3D1
  Cmax will define Tmax (time at wich Cmax is observed). For each time frame: at pre-dose of both study drugs and at 1, 2, 4 and 6 hours post- Pexidartinib dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - IUCT-oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voissiere A, Gomez-Roca C, Chabaud S, Rodriguez C, Nkodia A, Berthet J, Montane L, Bidaux AS, Treilleux I, Eberst L, Terret C, Korakis I, Garin G, Perol D, Delord JP, Caux C, Dubois B, Menetrier-Caux C, Bendriss-Vermare N, Cassier PA. The CSF-1R inhibitor pexidartinib affects FLT3-dependent DC differentiation and may antagonize durvalumab effect in patients with advanced cancers. Sci Transl Med. 2024 Jan 24;16(731):eadd1834. doi: 10.1126/scitranslmed.add1834. Epub 2024 Jan 24. PMID 38266104